CLINICAL TRIAL: NCT00523913
Title: Clinical Evaluation of Rosiglitazone Malate (BRL49653C) in Patients With Type 2 Diabetes Mellitus -Long-term Study of Rosiglitazone Maleate-
Brief Title: A Study Of BRL49653C For The Treatment Of Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVD105720
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes mellitus;; diabetes;; rosiglitazone; Avandia;
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rosiglitazone

SUMMARY:
This study is designed to evaluate the safety of BRL49653C administrated for 52 weeks

ELIGIBILITY:
Inclusion Criteria:

- Patients with type 2 diabetes mellitus managed by diet therapy or one antidiabetic agent (sulfonylurea or alpha glucosidase inhibitor) will be candidates for this study. These candidates will be checked up on their clinical laboratory data, and must have adequate blood, liver and kidney function.

Exclusion Criteria:

- Patient with serious cardiovascular disease or serious hepatic disease will not be eligible.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-11; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The safety profile (adverse events, laboratory parameters and other observations) of BRL49653C administered for 52 weeks will be evaluated. | 52 Weeks

SECONDARY OUTCOMES:
The efficacy profile (HbA1c, FPG and Insulin) of BRL49653C administered for 52 weeks will be evaluated. | 52 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: AVD105720 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AVD105720 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AVD105720 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AVD105720 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVD105720 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AVD105720 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AVD105720 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register